CLINICAL TRIAL: NCT05756348
Title: An Evaluation of the Skin Protection Characteristics of Two Commercially Available Skin Barrier Protectants
Brief Title: Durability of Two Skin Barrier Protectants (SBP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MED-2022-DIV71-003
Record Dates: First submitted 2022-10-19; First posted 2023-03-06 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-08

CONDITIONS: Skin Hydration in Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- receives both product (Other): all participants receive both products under evaluation.
  Interventions: Device: Marathon® XL No Sting Cyanoacrylate Skin Protectant and 3M™ Cavilon™ Advanced Skin Protectant

INTERVENTIONS:
Device: Marathon® XL No Sting Cyanoacrylate Skin Protectant and 3M™ Cavilon™ Advanced Skin Protectant — All participants will receive both device interventions listed above.

SUMMARY:
The current study will evaluate the duration of wear and durability of two commercially available SBPs: Medline Marathon® XL (extra long) No Sting Cyanoacrylate Skin Protectant (henceforth referred to as "Marathon®") and 3M™ Cavilon™ Advanced Skin Protectant (henceforth referred to as "Cavilon™").

DETAILED DESCRIPTION:
Completion of informed consent and participant screening will be followed by a washout period of minimum 18 hours (wherein participants will be asked to avoid application of cleansers, lotions, or perfumes to both forearms and inner elbows) prior to the first visit (Visit 1) of the study. During Visit 1, study personnel will confirm that the washout period has been successfully completed. Participants will wash their forearms and inner elbows with a standardized soap and dry them using paper towels for each arm. After the participants' forearms and inner elbows have fully dried, study personnel will use a Corneometer® (which measures skin hydration) to record baseline measurements of the skin within 2-inch x 2-inch squares (starting about two inches above the wrist) marked with a non-toxic marker on the volar forearms and inner elbows of the participants. Thereafter, participants will be randomized to the two SBPs, Marathon® or Cavilon™ (designated SBP). The designated SBP will be applied to the volar forearm and inner elbow "test areas" on the participant's dominant arm (as determined by the participant). The other SBP will be applied to the volar forearm and inner elbow "test areas" on the participant's non-dominant arm. A distinct area of each volar forearm will be used as an "untreated control area". Corneometer® measurements will be taken again on the same day after the SBPs have been left to dry for at least one minute or have fully dried. Thereafter, subsequent measurements will be taken daily over a seven-day period with a two-day break over the weekend. Each participant will commence the study on Monday or Tuesday. This will permit daily readings for the first 72 hours, which is the more important window to evaluate SBP wear time. There will be a two-day break in measurements over the weekend, after which Corneometer® measurements will be taken either on Monday, or Monday and Tuesday, depending on the participants' start date. Participants will be allowed to bathe their arms using a standardized soap provided by the study personnel but will be asked to minimize scrubbing and any other abrasion of the volar forearms and inner elbows. In addition, participants will be instructed not to engage in activities, for eg, sports (eg, tennis) or holding a baby that may cause significant abrasion on one arm and not the other. On the last visit of the study (Visit 6), study personnel will take the last set of Corneometer® measurements. In addition, participants will also complete surveys regarding their experience with the SBPs on specific days during study participation.

The Corneometer® measurements will help determine the presence of the SBPs and their deterioration over time. Skin treated with the SBPs will typically have lower readings than untreated skin. As the SBPs break down, the corresponding readings are expected to rise.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age

Exclusion Criteria:

* Individuals have skin conditions that might interfere with Corneometer® measurements, including rash, irritation, sunburn, tattoo, birthmark, any other dermal irregularities on the left or right volar forearm or inner elbow.
* Individuals have excessive hair on the left or right volar forearm or inner elbow as determined by study personnel.
* Individuals have a self-reported allergy/sensitivity to ingredients present in either of the SBPs, components of the soap used for bathing, or the exam gloves and non-toxic marker used in the study.
* Individuals are pregnant.
* Individuals whose self-reported activities may affect friction on one arm more than the other (eg, sports like tennis or holding a baby where one arm is used more routinely than the other).
* Individuals who are able to identify the manufacturer of the SBPs included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Miller, Principal Investigator — Medline Industries, LP
Locations (1):
- Medline Industries, LP, Northfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received both the Medline and Cavilon products. Analysis was performed per product not per arm randomization. The dominant arm of participants was randomized to receive one intervention (i.e., " Marathon® or Cavilon™ ), and the non-dominant arm received the other intervention.
Units Other Than Participants: arms
Groups:
- All Participants: all participants receive both products under evaluation.
  Marathon® XL No Sting Cyanoacrylate Skin Protectant and 3M™ Cavilon™ Advanced Skin Protectant: All participants will receive both device interventions listed above.
Period: Overall Study
Arm/Group | All Participants
Started | 42; 84 arms
Received Marathon | 42; 42 arms
Received Cavilon | 42; 42 arms
Completed | 42; 84 arms
Not Completed | 0; 0 arms

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 20
  Female | 21
  Other | 0
  Decline to Answer | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fitzpatrick Skin Assessment Scale [Count of Participants; unit: Participants]
  I (very fair) | 1
  II (fair) | 15
  III (medium) | 20
  IV (olive) | 5
  V (brown) | 1
  VI (dark brown) | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration
Description: To evaluate the duration of wear of Marathon® and Cavilon™ using the Corneometer® CM (capacitance method) 825 taking measurements of the skin (in Arbitrary Units) with the skin protectant applied at various time points compared to the skin control site without skin protectant at the same time points.
Time Frame: 7 Days - Baseline + 6 visits = 7
Population: Low arbitrary units correlate with less moisture (better skin protectant). As skin protectant wears off, arbitrary units will increase over time indicating duration of wear of skin protectant.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- All Participants: all participants received both products
Arm/Group | All Participants
Number analyzed (Participants) | 42
arbitrary units
  Marathon Baseline 0 | 36.71 (9.99)
  Cavilon Baseline 0 | 36.31 (1.6)
  Marathon Follow-up 1 | 7.95 (5.31)
  Cavilon Follow-up 1 | 20.98 (1.34)
  Marathon Follow-up 2 | 9.58 (7.80)
  Cavilon Follow-up 2 | 17.00 (6.06)
  Marathon Follow-up 3 | 15.71 (7.73)
  Cavilon Follow-up 3 | 17.67 (5.68)
  Marathon Follow-up 4 | 20.23 (9.18)
  Cavilon Follow-up 4 | 19.2 (7.82)
  Marathon Follow-up 5 | 23.07 (10.66)
  Cavilon Follow-up 5 | 22.51 (9.16)
  MarathonFollow-up 6 | 26.99 (8.82)
  Cavilon Follow-up 6 | 23.96 (10.06)

2. Primary Outcome: Durability
Description: To evaluate the durability of Marathon® and Cavilon™ using the Corneometer® CM 825 taking measurements of the skin (in Arbitrary Units) in the inner elbow location with the skin protectant applied at various time points compared to the skin control site without skin protectant at the same time points.
Time Frame: 7 Days - Baseline + 6 visits = 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Receives Both Product
Number analyzed (Participants) | 42
percent change
  Marathon Visit 0 | 3.00 (4.33)
  Cavilon Visit 0 | 4.49 (6.14)
  Marathon Visit 1 | 1.37 (5.11)
  Cavilon Visit 1 | 2.70 (6.01)
  Marathon Visit 2 | -0.59 (4.11)
  Cavilon Visit 2 | 2.53 (5.93)
  Marathon Visit 3 | 2.10 (5.27)
  Cavilon Visit 3 | 2.65 (4.68)
  Marathon Visit 4 | 5.10 (6.71)
  Cavilon Visit 4 | 2.72 (6.23)
  Marathon Visit 5 | 7.21 (7.45)
  Cavilon Visit 5 | 2.32 (6.86)
  Marathon Visit 6 | 8.50 (7.02)
  Cavilon Visit 6 | 4.25 (6.46)

3. Secondary Outcome: Participant Feedback 2
Description: To collect information on the participant experience with the two SBPs (Skin Barrier Protectants) using survey results (5 point scale from very comfortable to very uncomfortable). This question was on assessed at visit one.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Receives Both Product
Number analyzed (Participants) | 42
Participants
  Marathon Visit 1: Is the SBP comfortable on your arm: Very Comfortable | 3
  Marathon Visit 1: Is the SBP comfortable on your arm: Comfortable | 10
  Marathon Visit 1: Is the SBP comfortable on your arm: Neutral | 11
  Marathon Visit 1: Is the SBP comfortable on your arm: Uncomfortable | 18
  Marathon Visit 1: Is the SBP comfortable on your arm: Very Uncomfortable | 0
  Cavilon Visit 1: Is the SBP comfortable on your arm: Very Comfortable | 8
  Cavilon Visit 1: Is the SBP comfortable on your arm: Comfortable | 25
  Cavilon Visit 1: Is the SBP comfortable on your arm: Neutral | 6
  Cavilon Visit 1: Is the SBP comfortable on your arm: Uncomfortable | 2
  Cavilon Visit 1: Is the SBP comfortable on your arm: Very Uncomfortable | 1

4. Secondary Outcome: Participant Feedback
Description: To collect information on the participant experience with the two SBPs using survey results (yes/no questions). This measurement collected on visit thee and visit six.
Time Frame: 2 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Receives Both Product
Number analyzed (Participants) | 42
Participants
  Marathon Visit 3: Do you see the SBP on your skin?: yes | 36
  Marathon Visit 3: Do you see the SBP on your skin?: no | 6
  Cavilon Visit 3: Do you see the SBP on your skin?: yes | 37
  Cavilon Visit 3: Do you see the SBP on your skin?: no | 5
  Marathon Visit 3: Did the SBP accumulate dirt or debris?: yes | 10
  Marathon Visit 3: Did the SBP accumulate dirt or debris?: no | 32
  Cavilon Visit 3: Did the SBP accumulate dirt or debris?: yes | 20
  Cavilon Visit 3: Did the SBP accumulate dirt or debris?: no | 22
  Marathon Visit 3: Did the SBP adhere to clothing or material?: yes | 8
  Marathon Visit 3: Did the SBP adhere to clothing or material?: no | 34
  Cavilon Visit 3: Did the SBP adhere to clothing or material?: yes | 19
  Cavilon Visit 3: Did the SBP adhere to clothing or material?: no | 23
  Marathon Visit 6: Do you see the SBP on your skin?: yes | 37
  Marathon Visit 6: Do you see the SBP on your skin?: no | 5
  Cavilon Visit 6: Do you see the SBP on your skin?: yes | 36
  Cavilon Visit 6: Do you see the SBP on your skin?: no | 6
  Marathon Visit 6: Did the SBP accumulate dirt or debris?: yes | 10
  Marathon Visit 6: Did the SBP accumulate dirt or debris?: no | 32
  Cavilon Visit 6: Did the SBP accumulate dirt or debris?: yes | 20
  Cavilon Visit 6: Did the SBP accumulate dirt or debris?: no | 22
  Marathon Visit 6: Did the SBP adhere to clothing or material?: yes | 8
  Marathon Visit 6: Did the SBP adhere to clothing or material?: no | 34
  Cavilon Visit 6: Did the SBP adhere to clothing or material?: yes | 19
  Cavilon Visit 6: Did the SBP adhere to clothing or material?: no | 23

5. Secondary Outcome: Participant Feedback - Product Preference
Description: Collect participant feedback on which arm is it easier to determine the skin barrier protectant is present?
Time Frame: 7 Days - Baseline + 6 visits = 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 42
Participants
  Marathon | 7
  Cavilon | 35

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Marathon® XL No Sting Cyanoacrylate Skin Protectant; 3M™ Cavilon™ Advanced Skin Protectant: all participants receive both products under evaluation, however, clinical trials.gov requested adverse events be reported as separate arms per intervention.
Arm/Group | Marathon® XL No Sting Cyanoacrylate Skin Protectant | 3M™ Cavilon™ Advanced Skin Protectant
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT05756348/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05756348/ICF_001.pdf